CLINICAL TRIAL: NCT00565214
Title: Effect of Supplementary Vitamins on Oxidant Gene Expression in the Lungs of Healthy Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 0705009179
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: vitamin supplements; healthy smokers; epithelial lung tissue; bronchoscopy; antioxidant levels
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ascorbic Acid; Vitamin E; Selenium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): On Day 1, Group 1 will initiate in a double-blinded fashion, a once daily vitamin combination of selenomethionine(400 μg), vitamin E(400 IU), and vitamin C (1000 mg) orally for 30 days at home. After 30 days of treatment with Vitamin supplements, the gene expression of the airway epithelium will be compared to that of the Placebo group.
  Interventions: Dietary Supplement: Group 1
- Group 2 (Placebo Comparator): On Day 1, Group 2 will initiate the placebo in a double-blinded fashion.
  Interventions: Dietary Supplement: Group 2

INTERVENTIONS:
Dietary Supplement: Group 1 — The treatment plan involves the administration of a combination of 3 vitamins (vitamin C 1000 mg, vitamin E 400 IU, selenomethionine 400 μg) to study volunteers in a 2:1 randomization, Vitamins are to be taken orally, once a day, for a duration of 30 days.
  Other Names: Vitamin C, Vitamin E, Selenium
  Arms: Group 1
Dietary Supplement: Group 2 — The treatment plan involves the administration of a combination of 3 placebos to be taken orally, once daily for a duration of 30 days.
  Other Names: Placebo
  Arms: Group 2

SUMMARY:
Smoking damages the airway epithelium. The major mechanism by which this is done is by molecules called free radicals. Our body attempts to deal with these damaging molecules in two ways. One mechanism is via the presence of protective anti-oxidant vitamins and the other is via proteins that are produced by the body to convert free radicals to safer, less reactive molecules. Vitamins in our diet play a significant role in antioxidant defenses by directly neutralizing the damaging free-radicals and by providing co-factors to cellular proteins that neutralize the free radicals. This project is designed to look at the effects of giving individuals supplemental vitamins to see if it improves their defenses against oxidant insults. The investigators plan to look at the effects of these supplements over a 30 day period and monitor the effects by measuring vitamin levels in the blood and in the lung, and by measuring the response of cells in the lung through the increase or decrease in expression of genes responsive to oxidants.

To participate in this protocol, the research subject should first be enrolled in Weill-IRB protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy", fulfilling the inclusion/exclusion criteria of that protocol. They will be invited to participate in this Vitamin protocol only if they meet the additional inclusion/exclusion criteria of this protocol.

DETAILED DESCRIPTION:
The purpose of this study is to test whether dietary antioxidant supplementation can alter the expression in lung epithelial cells of genes related to oxidant response and whether this response is dependent on factors such as the individual's baseline serum antioxidant status, dietary antioxidant status, and the oxidant/anti-oxidant balance in the lung. The underlying hypothesis is that the intake of vitamins with antioxidant properties (selenomethionine, vitamin E and vitamin C) will boost the antioxidant levels of the airway epithelium sufficient to protect the epithelium from the stress of oxidants in cigarette smoke. Our prior work shows that phenotypic normal smokers (cigarette smokers with normal history, physical exam, lung function tests, and chest x-rays) have marked up and down regulation of > ~200 genes in the airway epithelium. The proposed project will build on past findings by examining whether regulation of gene expression responds to changes in nutritional status. The primary aim will be assessment of gene expression of the airway epithelium (from protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy") obtained before and after taking standard amounts of selenomethionine, vitamin E and vitamin C, or placebo for 30 days. The secondary aims will be to evaluate the ability of vitamin supplementation to raise lung and serum vitamin levels, to reduce the oxidant stress in the lung and systemically (as measured by lung and urinary F2 isoprostane levels, respectively), and to assess the vitamin-induced change in airway epithelial gene expression in genes other than oxidant related genes.

ELIGIBILITY:
Inclusion Criteria:

* All study individual should be enrolled in Weill-IRB protocol #0005004439 entitled "Evaluation of the Lungs of Normal (Smokers, Ex-smokers, Non-Smokers) Individuals with Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing, and Bronchial Wall Biopsy."
* All study subjects should be able to provide informed consent.
* Males or females ages 18 years and older.
* Current smokers with at least a 15 pack-year history (1 pack year = on average 20 cigarettes per day for 1 year).

Exclusion Criteria:

* Drug and/or alcohol abuse within the past six months.
* Individuals already on supplemental vitamins.
* Subjects intending to quit smoking in the next 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The effects of the supplements on gene expression | After 30 days of intervention
  To test whether 1 month of dietary antioxidant vitamin supplements alter the expression in lung epithelial cells of genes related to oxidant response.

SECONDARY OUTCOMES:
Vitamin supplementation | After 30 days of intervention
  The ability of vitamin supplementation to raise lung and serum vitamin levels will be evaluated.
Oxidant stress in the lung. | After 30 days of intervention
  The levels of oxidant stress in the lung will be evaluated.
Changes in airway epithelial gene expression in genes other than oxidant related genes. | After 30 days of intervention
  To determine whether the vitamin supplementation can induce changes in airway epithelial gene expression in genes other than oxidant related genes.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided